CLINICAL TRIAL: NCT00634491
Title: Effect of Acetazolamide in Prevention of Contrast Nephropathy
Brief Title: Comparison Between Effect of Acetazolamide and NaHco3 in Prevention of Contrast Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Fars Heart Foundation (Unknown)
Responsible Party: Office of Vice Chancellor for research in Shiraz UMS, Shiraz University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2438
Record Dates: First submitted 2008-02-14; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Contrast Induced Nephropathy
MeSH Terms: interventions — Sodium Bicarbonate; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 150 meq/l NaHco3 3cc/kg/hr one Hour before and 1cc/kg/hr 6 hour after angiography
  Interventions: Drug: sodium bicarbonate
- 2 (Active Comparator): Acetazolamide 250 mg + 1cc/kg/hr normal salin 6 hour before and after angiography
  Interventions: Drug: Acetazolamide
- 3 (Active Comparator): normal salin 1cc/kg/hr before and after angiography
  Interventions: Drug: normal salin

INTERVENTIONS:
Drug: sodium bicarbonate — 150 meq/l Sodium bicarbonate 3cc/kg/hr before and 1cc/kg/hr after angiography
  Other Names: no other name
  Arms: 1
Drug: Acetazolamide — Acetazolamide 250 mg+ 1 cc/kg/hr normal salin before and after angiography
  Other Names: Diamox
  Arms: 2
Drug: normal salin — 1 cc/kg/hr 6 hour before and after angiography
  Other Names: no other name
  Arms: 3

SUMMARY:
The purpose of this study is whether Acetazolamide is effective in prevention of contrast nephropathy

DETAILED DESCRIPTION:
Contrast induced nephropathy is one of common causes of acute renal failure many preventive protocol existed . 240 patient that underwent coronary angiography randomly divided in three groups.Group 1,2,3 will receive Bicarbonate ,Acetazolamide+Normal salin and Normal salin respectively.We compare prevalence of contrast nephropathy in each group.

ELIGIBILITY:
Inclusion Criteria:

* patient that underwent coronary angiography

Exclusion Criteria:

* serum Cr. more than 3 mg/dl
* electrolyte and acid-base imbalance
* pulmonary edema
* allergy to Acetazolamide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Increased base line creatinine at least 25% | 24 hr later

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Pakfetrat, MD, Study Chair — Shiraz nephro-urology research center
Locations (1):
- Fars Heart Foundation , Kowsar hospital, Shiraz, Iran

REFERENCES:
- [Result] Assadi F. Acetazolamide for prevention of contrast-induced nephropathy: a new use for an old drug. Pediatr Cardiol. 2006 Mar-Apr;27(2):238-42. doi: 10.1007/s00246-005-1132-z. PMID 16391986